CLINICAL TRIAL: NCT01028300
Title: Clinical Outcomes of Lumbar Degenerative Disc Disease Treated Operatively in Active-Duty U.S. Service Personnel With Lumbar Total Disc Replacement
Brief Title: Clinical Outcomes of Lumbar Degenerative Disc Disease in Active-Duty U.S. Service Personnel
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to enrollment failure
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Military ProDisc-L Study
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Degenerative Disc Disease
Keywords: DDD
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ProDisc L (Other)
  Interventions: Device: ProDisc™-L Total Disc Replacement (TDR)

INTERVENTIONS:
Device: ProDisc™-L Total Disc Replacement (TDR) — The design is based on a ball and socket articulation, one surface being metal and the other an ultra-high molecular weight polyethylene (UHMWPE). Three components comprise this modular prosthesis.

SUMMARY:
Degenerative disc disease (DDD) refers to a syndrome in which a degenerating disc causes chronic back pain, significantly impacting an individual's ability to function. The condition is most commonly diagnosed in the lumbosacral spinal segments L3-S1. The condition often starts with an injury to the disc space. The injury weakens the disc and creates excessive motion at the corresponding vertebral level. Over time, the segmental instability and associated neurological compromise combined with ongoing inflammatory processes that occur in and around the disc produce low back pain. The reparative processes in the disc are poor, thus the painful symptoms can become chronic.

Premature degeneration at adjacent levels of the spine remains one of the more vexing problems facing spinal surgeons when advising relatively young people to consider lumbar fusion surgery. Stopping the motion changes the mechanics of the back (which is designed for motion and flexibility) and results in the transfer of the loads and stresses to the adjacent vertebral segments. It is therefore intuitive to pursue total disc replacement, which allows for the treatment of pain due to DDD while re-establishing motion and stability, load distribution, and restoring the disc height, as an alternative to spinal fusion surgery.

The study hypothesis is that military personnel receiving Total Disc Replacement will return to the same level of active duty performance as at the time of their most recent successful physical readiness test.

ELIGIBILITY:
Inclusion Criteria:

1. Degenerative Disc Disease (DDD) in one vertebral level between L3 and S1, where a diagnosis of DDD requires:

   1. Back and/or leg (radicular) pain; and
   2. Radiographic confirmation of any one of the following by CT, MRI, discography, plain film, myelography, and/or flexion/extension films:

   i. Decreased disc height > 2 mm; ii. Scarring/thickening of annulus fibrosis; iii. Herniated nucleus pulposus; or iv. Vacuum phenomenon.
2. Skeletally mature adult between the ages of 18 and 50 years at time of surgery.
3. Failed at least 6 months of conservative therapy.
4. Oswestry Low Back Pain Disability Questionnaire score ≥ 20/50 (40%) (Interpreted as moderate/severe disability).
5. Psychosocially, mentally and physically able to fully comply with this protocol including adhering to scheduled visits, treatment plan, completing forms, and other study procedures.
6. Plans to remain on active duty for a minimum of two (2) years.
7. Personally signed and dated the informed consent document prior to any study-related procures indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. More than one vertebral level to be treated.
2. The involved vertebral endplates dimensionally smaller than 34.5 mm in the medial-lateral direction and/or 27 mm in the anterior-posterior direction.
3. Known allergy to polyethylene, cobalt chromium, or molybdenum
4. Prior fusion surgery at any lumbar vertebral level.
5. Clinically compromised vertebral body at the affected level due to current or past trauma.
6. Radiographic confirmation of facet joint disease or degeneration.
7. Lytic spondylolisthesis or spinal stenosis.
8. Degenerative spondylolisthesis > Grade 1.
9. Osteoporosis: A screening questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation), will be used to screen patients who require a DEXA bone mineral density measurement. If DEXA is required, exclusion will be defined as a DEXA bone density measured T score </= -2.5.
10. Known history of Paget's disease, osteomalacia, or any other metabolic bone disease.
11. Morbid obesity defined as a body mass index > 40 kg/m2 or weight more than 100 pounds over ideal body weight.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center - San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ProDisc L
Started | 4
Completed | 0
Not Completed | 4
Not completed — Study Terminated | 4

BASELINE CHARACTERISTICS:
Arm/Group | ProDisc L
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study is the Assessment of the Mean Oswestry Low Back Pain Disability Questionnaire (ODI) Improvement at the Twelve (12) Month and Twenty-four (24) Month Follow-up Visits Relative to Baseline.
Time Frame: 24 months
Population: Study was terminated early due to slow enrollment. 1 subject was enrolled but not treated due to study termination. 1 subject was enrolled and treated, but had no follow-up visits due to study termination. Only Two subjects were seen for follow-up visits, and only at 3 months post surgery.
Arm/Group | ProDisc L
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Return to Active Duty
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | ProDisc L
Number analyzed (Participants) | 0

3. Secondary Outcome: No Re-operations, Revisions, Removals or Supplemental Fixation
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | ProDisc L
Number analyzed (Participants) | 0

4. Secondary Outcome: No Implant Related Complications
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | ProDisc L
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 and 24 months
Arm/Group | ProDisc L
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProDisc L (N=4)
Non-infected seroma (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ProDisc L (N=4)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Emesis (Gastrointestinal disorders) | 1 (1)
Pain-abdomen (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early due to slow enrollment. Only Two subjects were seen for follow-up visits, and only at 3 months post surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Investigators may freely present or publish results of the Clinical Investigation in a manner which fairly sets forth the conclusions reached by the Clinical Investigators, but only after the Sponsor has been given the opportunity of reviewing the proposed presentation or publication prior to the intended submission, presentation, or publication date